CLINICAL TRIAL: NCT03026933
Title: A Multi-center, Randomized, Double Blind, Parallel Phase III Study to Evaluate the Efficacy and Safety of KI1107 in Patients Whose TG Level is Not Adequately Controlled With Rosuvastatin Calcium Monotherapy While LDL-C is Properly Controlled
Brief Title: Evaluate the Efficacy and Safety of KI1107 in Patients Whose TG Level is Not Adequately Controlled With Rosuvastatin Calcium Monotherapy While LDL-C is Properly Controlled
Acronym: ROMANTIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-OR-8301
Record Dates: First submitted 2017-01-16; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): KI1107
  Interventions: Drug: KI1107 4 Capsules, QD
- Control (Active Comparator): Rosuvastatin calcium
  Interventions: Drug: Rosuvastatin Calcium 20 MG, QD

INTERVENTIONS:
Drug: KI1107 4 Capsules, QD — KI1107 4 Capsules
  Arms: Treatment
Drug: Rosuvastatin Calcium 20 MG, QD — Rosuvastatin Calcium 20mg, QD
  Arms: Control

SUMMARY:
To examine variation rate of Non-HDL with KI1107 comparison Rosuvastatin monotherapy.

DETAILED DESCRIPTION:
Study design:

Randomly assigned to two groups(KI1107 or Rosuvastatin monotherpy) after 4 weeks run-in period and prescribed KI1107 or Rosuvastatin for 8 weeks.

ELIGIBILITY:
Inclusion criteria:

* Screening Visit

  * Age: 19-80
  * High risk for cardiovascular disease according to NCEP APT III
  * TG≥130mg/dL and 160mg/dL>LDL-C≥100mg/dL for subjects who were not taking statins for 4 weeks
  * 500mg/dL>TG≥200mg/dL and LDL-C<110mg/dL for subjects who were taking statins for 4 weeks
* Baseline Visit

  * 500mg/dL>TG≥200mg/dL
  * LDL-C<110mg/dL
  * Reduction of LDL-C dompairng screening visit

Exclusion criteria:

* The patient has histories of acute artery disease within 3 months
* The patient has histories of operation revasculatiation or aneurysm within 6 months
* The patient has histories of Unexplained myaliga or diagnosed myalgia or rhabdomyolysis
* The patient has histories of Effectable disease to the procedrue and clinical trial result

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Variation rate of Non HDL-C | 8 weeks

SECONDARY OUTCOMES:
Variation rate of TG | 4 weeks, 8 weeks
Variation rate of Non HDL-C | 4 weeks
Variation rate of TC | 4 weeks, 8 weeks
Variation rate of LDL-C | 4 weeks, 8 weeks
Variation rate of VLDL-C | 4 weeks, 8 weeks
Variation rate of Apo A-I | 4 weeks, 8 weeks
Variation rate of Apo B | 4 weeks, 8 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim CH, Han KA, Yu J, Lee SH, Jeon HK, Kim SH, Kim SY, Han KH, Won K, Kim DB, Lee KJ, Min K, Byun DW, Lim SW, Ahn CW, Kim S, Hong YJ, Sung J, Hur SH, Hong SJ, Lim HS, Park IB, Kim IJ, Lee H, Kim HS. Efficacy and Safety of Adding Omega-3 Fatty Acids in Statin-treated Patients with Residual Hypertriglyceridemia: ROMANTIC (Rosuvastatin-OMAcor iN residual hyperTrIglyCeridemia), a Randomized, Double-blind, and Placebo-controlled Trial. Clin Ther. 2018 Jan;40(1):83-94. doi: 10.1016/j.clinthera.2017.11.007. Epub 2017 Dec 7. PMID 29223557